CLINICAL TRIAL: NCT01259986
Title: Treatment of Recalcitrant Forms of Vitiligo With a Low-energy 635 nm Visible Light Laser
Brief Title: Treatment of Vitiligo With Low-energy Visible Light Laser
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 3 patients enrolled, no meaningful repigmentation observed. Recruitment halted.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB6452
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Vitiligo
Keywords: Vitiligo; Laser; Segmental vitiligo; Acral vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser treatment (Experimental)
  Interventions: Procedure: Laser treatment

INTERVENTIONS:
Procedure: Laser treatment — Laser treatment of using 635 nm laser with a dose of 3.0 J/cm^2 to small area (2cm x 2cm) of vitiligo once to twice a week for a total of 12 weeks.

SUMMARY:
The purpose of this study is the evaluate the efficacy of using a low-energy 635 nm visible light laser in the treatment of various recalcitrant forms of vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a pigmentary disorder characterized by depigmented and hypopigmented macules and patches. There are forms of vitiligo which are more resistant to treatment, including segmental vitiligo and acral vitiligo. Previous studies have shown that a low energy helium-neon (633 nm) laser can cause increased proliferation of melanocytes and repigmentation in segmental-type vitiligo. The goal of this study is to verify these results and show efficacy in other recalcitrant forms of vitiligo including acral vitiligo and post melanocyte-keratinocyte transplantation vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Have active or stable segmental vitiligo on the neck or face, acral vitiligo, or have undergone recent melanocyte-keratinocyte transplantation procedure (MKTP)
* Agree to abide by the Investigator's guidelines regarding photosensitizing drugs and photoprotection
* Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form
* Agree to follow and undergo all study-related procedures

Exclusion Criteria:

* Women who are lactating, pregnant, or planning to become pregnant
* Patients with a recent history of melasma, and other disorders of pigmentation with the exception of post inflammatory hyperpigmentation
* Patients with a known history of photosensitivity disorders
* Photosensitizing medications may be continued throughout of the study at the discretion of the investigator
* Patients with a known history of melanoma or non-melanoma skin cancers
* Concomitant use of tanning beds
* Any reason the investigator feels the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percent repigmentation | 24 clinic visits over 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H. Hamzavi, M.D., Principal Investigator — Henry Ford Health System